CLINICAL TRIAL: NCT01059799
Title: A Pan Asian Trial Comparing Efficacy and Safety of Insulin NN1250 and Insulin Glargine as Add on to OAD(s) in Subjects With Type 2 Diabetes (BEGIN™: ONCE ASIA)
Brief Title: Comparison of NN1250 Versus Insulin Glargine in Subjects With Type 2 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3586; U1111-1113-2441 (Other: WHO); JapicCTI-101039 (Registry Identifier: JAPIC)
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg OD (Experimental)
  Interventions: Drug: insulin degludec
- IGlar OD (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Insulin degludec injected subcutaneously (under the skin) once daily. The doses will be individually adjusted
  Arms: IDeg OD
Drug: insulin glargine — Insulin glargine injected subcutaneously (under the skin) once daily. The doses will be individually adjusted
  Arms: IGlar OD

SUMMARY:
This trial is conducted in Asia and Japan. The aim of this trial is to compare insulin degludec (NN1250) with insulin glargine both combined with oral antidiabetic drugs (OADs) in subjects with type 2 diabetes never treated with insulin.

ELIGIBILITY:
Inclusion Criteria:

* For Japan only: minimum age is 20 years
* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* Current treatment with monotherapy or combination of an insulin secretagouge (sulfonylurea or glinide) and metformin, with or without addition of alfa-glucosidase-inhibitors or a DPP-4 inhibitor with unchanged dosing for at least 3 months prior to visit 1. The dose(s) should as minimum be as stated: -Insulin secretagogue (sulfonylurea or glinide): Minimum half of the daily maximal dose according to local labelling -Metformin: alone or in combination (including fixed combination): Maximum tolerated dose - alfa-glucosidase-inhibitors: Minimum half of the daily maximal dose or maximum tolerated dose -DPP-4 (dipeptyl peptidase 4) inhibitor: According to local labelling
* HbA1c 7.0-10.0 % (both inclusive) by central laboratory analysis
* Body Mass Index (BMI) no higher than 35.0 kg/m^2

Exclusion Criteria:

* Use within the last 3 months prior to Visit 1 of: TZDs (thiazolidinediones), exenatide or liraglutide
* Cardiovascular disease, within the last 6 months prior to visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg)
* Pregnancy, breast-feeding, or the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements (for Thailand: adequate contraceptive measures are: diaphragm, condom (by the partner), intrauterine device in place for last three months before trial starts, sponge, cap with spermicide, contraceptive patch, approved hormonal implant (i.e. Norplant), oral contraceptives taken without difficulty for the last three months before trial starts, post menopausal state or sterilisation.)
* Cancer and medical history of cancer (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-12-16 (Actual); Study Completion 2010-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (41):
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Japan (12):
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Kamakura-shi, Kanagawa
  - Novo Nordisk Investigational Site, Kawasaki-shi
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hygo
  - Novo Nordisk Investigational Site, Ogawa
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Takatsuki-shi, Osaka
- Malaysia (7):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, George Town
  - Novo Nordisk Investigational Site, Georgetown, Penang
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Kuala Selangor
  - Novo Nordisk Investigational Site, Putrajaya
- South Korea (9):
  - Novo Nordisk Investigational Site, Bucheon-si
  - Novo Nordisk Investigational Site, Busan
  - Novo Nordisk Investigational Site, Goyang
  - Novo Nordisk Investigational Site, Incheon
  - Novo Nordisk Investigational Site, Jeonju
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon
  - Novo Nordisk Investigational Site, Wŏnju
  - Novo Nordisk Investigational Site, Yangsan
- Taiwan (7):
  - Novo Nordisk Investigational Site, Banqiao District
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Chiayi City
  - Novo Nordisk Investigational Site, Kaohsiung City
  - Novo Nordisk Investigational Site, Kaoshiung
  - Novo Nordisk Investigational Site, Taichung
  - Novo Nordisk Investigational Site, Taipei
- Thailand (5):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Bangkoknoi, Bangkok
  - Novo Nordisk Investigational Site, Chiang Mai
  - Novo Nordisk Investigational Site, Nakhon Ratchasima
  - Novo Nordisk Investigational Site, Songkhla

REFERENCES:
- [Background] Einhorn D, Handelsman Y, Bode BW, Endahl LA, Mersebach H, King AB. PATIENTS ACHIEVING GOOD GLYCEMIC CONTROL (HBA1c <7%) EXPERIENCE A LOWER RATE OF HYPOGLYCEMIA WITH INSULIN DEGLUDEC THAN WITH INSULIN GLARGINE: A META-ANALYSIS OF PHASE 3A TRIALS. Endocr Pract. 2015 Aug;21(8):917-26. doi: 10.4158/EP14523.OR. Epub 2015 Jun 29. PMID 26121451
- [Result] Ratner RE, Gough SC, Mathieu C, Del Prato S, Bode B, Mersebach H, Endahl L, Zinman B. Hypoglycaemia risk with insulin degludec compared with insulin glargine in type 2 and type 1 diabetes: a pre-planned meta-analysis of phase 3 trials. Diabetes Obes Metab. 2013 Feb;15(2):175-84. doi: 10.1111/dom.12032. Epub 2012 Dec 3. PMID 23130654
- [Result] Heller S, Mathieu C, Kapur R, Wolden ML, Zinman B. A meta-analysis of rate ratios for nocturnal confirmed hypoglycaemia with insulin degludec vs. insulin glargine using different definitions for hypoglycaemia. Diabet Med. 2016 Apr;33(4):478-87. doi: 10.1111/dme.13002. Epub 2015 Dec 13. PMID 26484727
- [Result] Sorli C, Warren M, Oyer D, Mersebach H, Johansen T, Gough SC. Elderly patients with diabetes experience a lower rate of nocturnal hypoglycaemia with insulin degludec than with insulin glargine: a meta-analysis of phase IIIa trials. Drugs Aging. 2013 Dec;30(12):1009-18. doi: 10.1007/s40266-013-0128-2. PMID 24170235
- [Result] Russell-Jones D, Gall MA, Niemeyer M, Diamant M, Del Prato S. Insulin degludec results in lower rates of nocturnal hypoglycaemia and fasting plasma glucose vs. insulin glargine: A meta-analysis of seven clinical trials. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):898-905. doi: 10.1016/j.numecd.2015.06.005. Epub 2015 Jun 18. PMID 26232910
- [Result] Vora J, Seufert J, Solberg H, Kinduryte O, Johansen T, Hollander P. Insulin degludec does not increase antibody formation versus insulin glargine: an evaluation of phase IIIa trials. Diabetes Obes Metab. 2016 Jul;18(7):716-20. doi: 10.1111/dom.12621. Epub 2016 Feb 8. PMID 26663320
- [Result] Vora J, Christensen T, Rana A, Bain SC. Insulin degludec versus insulin glargine in type 1 and type 2 diabetes mellitus: a meta-analysis of endpoints in phase 3a trials. Diabetes Ther. 2014 Dec;5(2):435-46. doi: 10.1007/s13300-014-0076-9. Epub 2014 Aug 1. PMID 25081590
- [Result] Aye MM, Atkin SL. Patient safety and minimizing risk with insulin administration - role of insulin degludec. Drug Healthc Patient Saf. 2014 Apr 30;6:55-67. doi: 10.2147/DHPS.S59566. eCollection 2014. PMID 24812526
- [Result] Onishi Y, Iwamoto Y, Yoo SJ, Clauson P, Tamer SC, Park S. Insulin degludec compared with insulin glargine in insulin-naive patients with type 2 diabetes: A 26-week, randomized, controlled, Pan-Asian, treat-to-target trial. J Diabetes Investig. 2013 Nov 27;4(6):605-12. doi: 10.1111/jdi.12102. Epub 2013 Jun 3. PMID 24843715
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 52 sites in 6 countries: Hong Kong (1), Japan (12), Malaysia (8), South Korea (19), Thailand (6) and Taiwan (6)
Pre-assignment Details: Subjects continued on their current treatment with oral antidiabetic drug(s) (OAD(s) treatment except for dipeptyl peptidase-4 (DPP-4) inhibitors, at the pre-randomisation dose level and dosing frequency.
Groups:
- IDeg OD: Insulin degludec (IDeg) was given once daily (OD) subcutaneously (under the skin) in the evening in combination with pre-trial OADs (except DPP-4 inhibitors) for 26 weeks. Insulin doses were individually adjusted.
- IGlar OD: Insulin glargine (IGlar) was given once daily (OD) subcutaneously (under the skin) according to approved labelling in combination with pre-trial OADs (except DPP-4 inhibitors) for 26 weeks. Insulin doses were individually adjusted.
Period: Overall Study
Arm/Group | IDeg OD | IGlar OD
Started | 289 | 146
Exposed | 284 (Five subjects withdrew before exposure to trial drug) | 146
Completed | 258 | 136
Not Completed | 31 | 10
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal criteria | 13 | 2
Not completed — Other | 12 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised subjects and missing data is imputed using last observation carried forward (LOCF).
  Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD | IGlar OD | Total
Number analyzed (Participants) | 289 | 146 | 435
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (9.8) | 58.1 (10.1) | 58.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 71 | 202
  Male | 158 | 75 | 233
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.4 (0.8) | 8.5 (0.8) | 8.5 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.4 (2.1) | 8.6 (1.9) | 8.5 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The Full analysis set (FAS) included all randomised subjects and missing data is imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 289 | 146
percentage of glycosylated haemoglobin | -1.24 (0.87) | -1.35 (0.87)

2. Secondary Outcome: Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The Safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 284 | 146
Episodes/100 years of patient exposure | 298 | 370

3. Secondary Outcome: Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of nocturnal confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The Safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 284 | 146
Episodes/100 years of patient exposure | 78 | 124

4. Secondary Outcome: Mean of 9-point Self Measured Plasma Glucose Profile (SMPG)
Description: Mean of SMPG after 26 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, before bedtime, at 4 am and before breakfast.
Time Frame: Week 26
Population: The FAS included all randomised subjects.The missing data is imputed using last observation carried forward (LOCF). For 25 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 270 | 140
mmol/L | 8.2 (1.8) | 8.0 (1.9)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 8/284 | 8/146
Other Adverse Events (participants affected / at risk) | 58/284 | 39/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=284) | IGlar OD (N=146)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ureteric calculus removal (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=284) | IGlar OD (N=146)
Diabetic retinopathy (Eye disorders) | 15 (16) | 6 (6)
Nasopharyngitis (Infections and infestations) | 26 (32) | 20 (26)
Upper respiratory tract infection (Infections and infestations) | 22 (29) | 16 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.